CLINICAL TRIAL: NCT03903796
Title: A Phase 3, Randomized, Multicenter, Double-blind, Double-dummy, Parallel-controlled Study to Evaluate the Safety and Efficacy of HS-10234 25 mg QD Versus TDF 300 mg QD for the Treatment of Patients With HBeAg+/- Chronic HBV Infection.
Brief Title: Study of the Efficacy and Safety of HS-10234 in Patients With Chronic Hepatitis B Virus Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-10234-301
Record Dates: First submitted 2019-03-03; First posted 2019-04-04 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Chronic HBV Infection
Keywords: HBeAg-positive or negative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HS-10234 25mg (Experimental): HS-10234 + TDF placebo for up to 96 weeks
  Interventions: Drug: HS-10234; Drug: TDF
- TDF 300mg (Active Comparator): TDF + HS-10234 placebo for up to 96 weeks
  Interventions: Drug: HS-10234; Drug: TDF
- Open-label HS-10234 (Experimental): All participants who complete the double-blind period (96 weeks) will be eligible to receive open-label HS-10234 until week 144 of the study.
  Interventions: Drug: HS-10234

INTERVENTIONS:
Drug: HS-10234 — Drug: HS-10234 HS-10234 25mg will administer orally once daily Drug: TDF placebo TDF placebo 300mg will administer orally once daily
Drug: TDF — Drug: TDF TDF 300mg will administer orally once daily Drug: HS-10234 placebo HS-10234 placebo 25mg will administer orally once daily
  Arms: HS-10234 25mg; TDF 300mg

SUMMARY:
The primary objective of this study is to compare the safety and efficacy of HS-10234 versus tenofovir disoproxil fumarate (TDF) in treatment-naive and treatment-experienced adults with chronic hepatitis B virus (HBV) infection.

DETAILED DESCRIPTION:
This is a phase 3, randomized, multicenter, double-blind, double-dummy, parallel-controlled, non-inferiority trial to evaluate the safety and efficacy of HS-10234 25 mg qd versus TDF 300 mg qd. Patients with chronic HBV infection who are positive or negative for the hepatitis B e antigen (HBeAg) will be randomly assigned (2:1) to receive either 25 mg HS-10234 or 300 mg TDF with matching placebo. Randomization will be done by a computer-generated allocation sequence stratified by plasma HBV DNA concentration (HBV DNA< 8 log10IU/mL；HBV DNA ≥8 log10IU/mL) and previous treatment experience (treatment-naive and treatment-experienced). All patients will receive 144 weeks of antiviral therapy. After 96 weeks of double-blind treatment, all subjects will be eligible to receive open-label HS-10234 until 144 weeks.

The primary efficacy endpoint is the proportion of patients with HBV DNA less than 20 IU/mL at week 48 in all patients who are randomly assigned and received at least one dose of study drug using a missing-equals-failed approach. Key pre-specified safety endpoints are bone and renal parameters at week 48. Other pre-specified endpoints include viral suppression, serologic response, normalization of alanine aminotransferase (ALT) levels and the emergence of resistance mutations at week 48, 96 and 144.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria to be eligible for participation in this study:

  1. Must have the ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study screening.
  2. Male and non-pregnant, non-lactating females, from 18 up to 65 years of age (based on the date of the screening visit). A negative serum pregnancy test at screening is required for female subjects of childbearing potential.
  3. Documented evidence of chronic HBV infection (e.g. HBsAg positive for more than 6 months).
  4. HBeAg-positive or HBeAg-negative chronic hepatitis B with all of the following: HBV DNA ≥ 2 x 104 IU/mL; Screening serum 1 ULN < ALT level ≤ 10 ULN.
  5. Treatment-naive subjects (defined as < 12 weeks of oral antiviral treatment with any nucleoside or nucleotide analogue) OR treatment-experienced subjects (defined as subjects meeting all entry criteria [including HBV DNA and serum ALT criteria] and with ≥ 12 weeks of previous treatment with any nucleoside or nucleotide analogue) will be eligible for enrollment. Treatment-experienced subjects receiving oral antiviral treatment at Screening must continue their treatment regimen until the time of randomization, when it will be discontinued.
  6. Any previous treatment with interferon (pegylated or non-pegylated) must have ended at least 6 months prior to the baseline visit.
  7. Estimated creatinine clearance (CLcr) ≥ 50 mL/min（using the Cockcroft-Gault method）based on serum creatinine and actual body weight as measured at the screening evaluation, as follows:

  （140-age in years）(body weight [kg]) (72)(serum creatinine [mg/dL]） 8) Normal ECG (or if abnormal, determined by the Investigator not to be clinically significant).

  9) Must be willing and able to comply with all study requirements.

Exclusion Criteria:

* Subjects who meet any of the following exclusion criteria are not to be enrolled in this study:

  1. Pregnant women, women who are breastfeeding or who believe they may wish to become pregnant during the course of the study.
  2. Males and females of reproductive potential who are unwilling to use an "effective", protocol specified method(s) of contraception during the study.
  3. Co-infection with HCV virus, HIV, or HDV.
  4. Evidence of hepatocellular carcinoma (e.g. as evidenced by recent imaging).
  5. Any history of, or current evidence of, clinical hepatic decompensation (e.g. ascites encephalopathy or variceal hemorrhage).
  6. Abnormal hematological and biochemical parameters, including:

     * Hemoglobin < 10 g/dl
     * Absolute neutrophil count < 0.75 × 109/L
     * Platelets ≤ 50 × 109/L
     * AST or ALT > 10 × ULN
     * Total Bilirubin > 2.5 × ULN
     * Albumin < 3.0 g/dL
     * INR > 1.5 × ULN (unless stable on anticoagulant regimen)
  7. Received solid organ or bone marrow transplant.
  8. Significant renal, cardiovascular, pulmonary, or neurological disease in the opinion of the investigator.
  9. Significant bone disease (e.g. osteomalacia, chronic osteomyelitis, osteogenesis imperfecta, osteochrondroses), or multiple bone fractures.
  10. Malignancy within the 5 years prior to screening, with the exception of specific cancers that are cured by surgical resection (basal cell skin cancer, etc).
  11. Currently receiving therapy with immunomodulators (e.g. corticosteroids), investigational agents, nephrotoxic agents, or agents capable of modifying renal excretion.
  12. Known hypersensitivity to study drugs, metabolites, or formulation excipients.
  13. Current alcohol or substance abuse judged by the investigator to potentially interfere with participant compliance.
  14. Any other clinical condition or prior therapy that, in the opinion of the Investigator, would make the subject unsuitable for the study or unable to comply with dosing requirements.
  15. Subjects on prohibited concomitant medications. Subjects on prohibited medications, otherwise eligible, will need a wash out period of at least 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 963 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Evaluation the percentage of Participants with Hepatitis B Virus (HBV) DNA < 20 IU/mL | Week 48
  The primary efficacy endpoint was the proportion of patients with HBV DNA < 20 IU/mL at week 48 in all patients who are randomly assigned and received HS-10234 25 mg or TDF 300 mg. The safety and tolerance were also observed in two treatment groups.

SECONDARY OUTCOMES:
Evaluation the percent Change from Baseline in Hip BMD | Week 48
  Percent Change from Baseline in Hip Bone Mineral Density (BMD) at Week 48
Evaluation the percent Change from Baseline in Spine BMD | Week 48
  Percent Change from Baseline in Spine BMD at Week 48
Evaluation the change from Baseline in Serum Creatinine | Week 48
  Change from Baseline in Serum Creatinine at Week 48

OTHER OUTCOMES:
Evaluation the proportion of Patients Achieving Hepatitis B Surface Antigen (HBsAg) Loss | Week 48, 96 and 144
  Proportion of Patients Achieving Hepatitis B Surface Antigen (HBsAg) Loss at Weeks 48, 96, 144
Evaluation the proportion of Patients Achieving HBsAg Seroconversion | Week 48, 96 and 144
  Proportion of Patients Achieving HBsAg Seroconversion at Weeks 48, 96, 144
Evaluation the proportion of patients achieving HBeAg loss | Week 48, 96 and 144
  Proportion of patients achieving HBeAg loss at weeks 48, 96, 144
Evaluation the proportion of patients achieving HBeAg seroconversion | Week 48, 96 and 144
  Proportion of patients achieving HBeAg seroconversion at weeks 48, 96, 144

CONTACTS AND LOCATIONS:
Overall Officials: Guo Xiaolin, MD, Principal Investigator — The First Hospital of Jilin University, Jilin Province
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

REFERENCES:
- [Derived] Liu ZH, Jin QL, Zhang YX, Gong GZ, Wu GC, Yao LF, Wen XF, Gao ZL, Huang Y, Yang DK, Chen EQ, Mao Q, Lin SD, Shang J, Gong HY, Zhong LH, Yin HF, Wang FM, Hu P, Zhang XQ, Gao QJ, Xia P, Li C, Niu JQ, Hou JL; TMF Study Group. [Safety profile of tenofovir amibufenamide therapy extension or switching in patients with chronic hepatitis B: a phase Ⅲ multicenter, randomized controlled trial]. Zhonghua Gan Zang Bing Za Zhi. 2024 Oct 20;32(10):893-903. doi: 10.3760/cma.j.cn501113-20240807-00366. Chinese. PMID 39528324
- [Derived] Liu ZH, Jin QL, Zhang YX, Gong GZ, Wu GC, Yao LF, Wen XF, Gao ZL, Huang Y, Yang DK, Chen EQ, Mao Q, Lin SD, Shang J, Gong HY, Zhong LH, Yin HF, Wang FM, Hu P, Zhang XQ, Gao QJ, Jin CN, Li C, Niu JQ, Hou JL; TMF Study Group. [Efficacy evaluation of extending or switching to tenofovir amibufenamide in patients with chronic hepatitis B: a phase Ⅲ randomized controlled study]. Zhonghua Gan Zang Bing Za Zhi. 2024 Oct 20;32(10):883-892. doi: 10.3760/cma.j.cn501113-20240807-00365. Chinese. PMID 39528323
- [Derived] Liu Z, Jin Q, Zhang Y, Gong G, Wu G, Yao L, Wen X, Gao Z, Huang Y, Yang D, Chen E, Mao Q, Lin S, Shang J, Gong H, Zhong L, Yin H, Wang F, Hu P, Wu Q, Pan C, Jia W, Li C, Sun C, Niu J, Hou J; TMF Study Group. 96-Week Treatment of Tenofovir Amibufenamide and Tenofovir Disoproxil Fumarate in Chronic Hepatitis B Patients. J Clin Transl Hepatol. 2023 Jun 28;11(3):649-660. doi: 10.14218/JCTH.2022.00058. Epub 2022 Nov 1. PMID 36969889
- [Derived] Liu Z, Jin Q, Zhang Y, Gong G, Wu G, Yao L, Wen X, Gao Z, Huang Y, Yang D, Chen E, Mao Q, Lin S, Shang J, Gong H, Zhong L, Yin H, Wang F, Hu P, Xiao L, Li C, Wu Q, Sun C, Niu J, Hou J; TMF Study Group. Randomised clinical trial: 48 weeks of treatment with tenofovir amibufenamide versus tenofovir disoproxil fumarate for patients with chronic hepatitis B. Aliment Pharmacol Ther. 2021 Nov;54(9):1134-1149. doi: 10.1111/apt.16611. Epub 2021 Sep 29. PMID 34587302